CLINICAL TRIAL: NCT00905255
Title: A Randomized, Open Label, Parallel-group (One-step Titration and Two-step Titration), Multicenter 52-Week Study Followed by a 24-Week Extension Assessing the Safety and Tolerability of AVE0010 Monotherapy in Patients With Type 2 Diabetes
Brief Title: GLP-1 Receptor Agonist Lixisenatide in Patients With Type 2 Diabetes for Glycemic Control and Safety Evaluation in Monotherapy (GETGOAL-MONO Japan LTS)
Acronym: GETGOAL-MONO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTS10888
Record Dates: First submitted 2009-05-14; First posted 2009-05-20 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: hyperglycemia; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — lixisenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide (Two-step Titration) (Experimental): 2-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector
- Lixisenatide (One-step Titration) (Experimental): 1-step initiation regimen of lixisenatide: 10 mcg QD for 2 weeks, then 20 mcg QD up to end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
Device: Pen auto-injector
  Other Names: OptiClik®

SUMMARY:
The purpose of this study is to compare the benefits and risks of lixisenatide (AVE0010) used as 2-step initiation regimen and 1-step initiation regimen in Japan, over a period of 24 weeks of treatment, followed by an extension up to Week 76.

The primary objective of this study is to evaluate the safety of lixisenatide once daily treatment in monotherapy at Week 24 by a descriptive comparison of a 1-step initiation and a 2-step initiation regimen in patients with type 2 diabetes in Japan.

The secondary objectives are to assess the overall safety of lixisenatide once daily treatment in monotherapy at Week 52 and Week 76; to assess the effects of lixisenatide on glycosylated hemoglobin (HbA1c) reduction at Week 52 and Week 76, body weight, and fasting plasma glucose (FPG); to assess pharmacokinetics (PK) and anti-lixisenatide antibody development.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed for at least 2 months at the time of screening visit, not treated by an antidiabetic agent in the 3 months before screening, except treatment with sulfonylureas or alpha-glucosidase inhibitors at a stable dose. In this case the oral antidiabetic treatment must be discontinued before starting single-blind run-in phase

Exclusion Criteria:

* HbA1c less than (<) 7 percent (%) or greater than (>) 10% at screening
* At the time of screening age <legal age of majority
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* Type 1 diabetes mellitus
* Type 2 diabetes treated by an antidiabetic pharmacological agent (except sulfonylurea or alpha-glucosidase inhibitors at a stable dose) within the 3 months preceding the screening. Insulin use is accepted if it is not within 3 months prior to screening visit and only for the following reasons: a) Prior insulin use for management of gestational diabetes; b) Short-term (less than or equal to [<=] 1 month) insulin use to maintain glycemic control for hospitalization, medical procedures, or intervention
* FPG at screening >250 milligram per deciliter (mg/dL) (>13.9 millimole per liter [mmol/L])
* Weight change of more than 5 kilogram (kg) during the 3 months preceding the screening visit
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within 3 months prior to the time of screening
* Within the last 6 months prior to screening: history of myocardial infarction, stroke, or heart failure requiring hospitalization
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting supine systolic or diastolic blood pressure >180 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Laboratory findings at the time of screening: aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP): >2 times upper limit of the normal (ULN) laboratory range; amylase and/or lipase: >3 times ULN; total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome); hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100000/mm^3; positive test for Hepatitis B surface antigen (HBsAg) and/or Hepatitis C antibody (HCAb) and positive serum pregnancy test in females of childbearing potential
* Any clinically significant abnormality identified on physical examination, laboratory tests, electrocardiogram (ECG) or vital signs at the time of screening that in the judgment of the investigator or any sub-investigator precludes safe completion of the study or constrains efficacy assessment
* Patients who are considered by the investigator or any sub-investigator as inappropriate for this study for any reason (for example, impossibility to meet specific protocol requirements, such as scheduled visits, being able to do self-injections, likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol)
* Patient is an investigator or any sub-investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to the time of screening
* Use of any investigational drug within 3 months prior to screening
* Participation in a previous study with lixisenatide
* End-stage renal disease as defined by a serum creatinine clearance of <15 milliliter/minute (calculated by the Cockcroft and Gault formula) and/or patients on dialysis
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to gastroparesis and gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening
* Allergic reaction to any glucagon like peptide-1 (GLP-1) agonist in the past (for example, exenatide, liraglutide) or to metacresol
* Additional exclusion criteria at the end of the run-in phase: informed consent withdrawal (patient not willing to continue or failed to return); lack of compliance during the single-blind placebo run-in phase (>2 injections missed); and patient with any adverse event which precludes the inclusion in the study, as assessed by the Investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan

REFERENCES:
- [Result] Seino Y, Yabe D, Takami A, Niemoeller E, Takagi H. Long-term safety of once-daily lixisenatide in Japanese patients with type 2 diabetes mellitus: GetGoal-Mono-Japan. J Diabetes Complications. 2015 Nov-Dec;29(8):1304-9. doi: 10.1016/j.jdiacomp.2015.07.003. Epub 2015 Jul 6. PMID 26342556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 centers in Japan between May 09, 2009 and January 22, 2011. The overall duration of treatment was at least 76 weeks (52-week open-label treatment; 24-week open-label extension treatment).
Pre-assignment Details: A total of 75 patients were screened of which 6(8.0%) were screen failures; main reasons for screen failure:glycosylated hemoglobin being out of defined protocol range (>=7% and <=10%) and use of an antidiabetic agent other than a sulfonylurea or alpha-glucosidase inhibitor within 3 months prior to screening. A total of 69 patients were randomized.
Groups:
- Lixisenatide (Two-step Titration): 2-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
- Lixisenatide (One-step Titration): 1-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 2 weeks, then 20 mcg QD up to end of treatment.
Period: Overall Study
Arm/Group | Lixisenatide (Two-step Titration) | Lixisenatide (One-step Titration)
Started | 33 (Randomized.) | 36
Safety Population | 33 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 36
Modified Intent-to-Treat(mITT)Population | 33 (All patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment.) | 36
Completed | 20 | 27
Not Completed | 13 | 9
Not completed — Adverse Event | 7 | 5
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Familial and Personal Reasons | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Lixisenatide (Two-step Titration): 2-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
- Total: Total of all reporting groups
Arm/Group | Lixisenatide (Two-step Titration) | Lixisenatide (One-step Titration) | Total
Number analyzed (Participants) | 33 | 36 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (9.0) | 60.4 (8.2) | 58.7 (8.7)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 30 | 28 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Asian/Oriental | 33 | 36 | 69
  Ethnicity: Non Hispanic | 33 | 36 | 69
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.35 (0.82) | 8.12 (0.68) | 8.23 (0.76)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 9.91 (1.91) | 9.16 (1.92) | 9.52 (1.94)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 70.75 (19.21) | 66.74 (11.14) | 68.66 (15.54)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated by dividing body weight by the height squared.
  kilogram per square meter (kg/m^2) | 25.16 (5.27) | 24.81 (3.68) | 24.98 (4.48)
Duration of Diabetes [Mean (Standard Deviation); unit: years] — Duration of diabetes is reported at screening.
  years | 8.05 (6.38) | 9.03 (7.87) | 8.56 (7.16)

OUTCOME MEASURES:

1. Secondary Outcome: Overview of Adverse Event Profile (Treatment Emergent Adverse Events) of All Patients During On-Treatment Period Assessed Through Adverse Events Collection and Vital Signs, ECG and Laboratory Monitoring
Description: Overview of adverse event profile is reported in terms of percentage of patients with TEAEs during the on-treatment period: any TEAE; any serious TEAE; any TEAE leading to death; any TEAE leading to permanent treatment discontinuation. The on-treatment period was the time from the first dose of study drug up to 3 days after the last dose at Week 76.
Time Frame: First dose of study drug up to 3 days after the last dose of study drug at Week 76 or early withdrawal
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered. Analysis was done on the overall group (pooled data from the 2-step and 1-step titration arms) as pre-specified
Measure: Number; unit: percentage of participants
Groups:
- Lixisenatide (Combined): Included all patients who received 2-step initiation regimen of lixisenatide or 1-step initiation regimen of lixisenatide.
Arm/Group | Lixisenatide (Combined)
Number analyzed (Participants) | 69
percentage of participants
  Any TEAE | 91.3
  Any Serious TEAE | 4.3
  Any TEAE Leading to Death | 0
  Any TEAE Leading to Treatment Discontinuation | 14.5

2. Other Pre Specified Outcome: Percentage of Patients Requiring Rescue Therapy
Description: Routine fasting self-monitored plasma glucose (SMPG) and central laboratory FPG (and HbA1c after Week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after Week 12) were performed. Threshold values - from Week 4 to Week 8: fasting SMPG/FPG >270 milligram/deciliter (mg/dL) (15.0 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8.5%, from Week 24 to end of treatment (Week 76): fasting SMPG/FPG >180 mg/dL (10.0 mmol/L) or HbA1c >8%. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 52, Baseline up to Week 76
Population: mITT population.Analysis was done on the overall group (pooled data from the 2-step and 1-step titration arms) as pre-specified
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide (Combined)
Number analyzed (Participants) | 69
percentage of participants
  Baseline up to Week 52 | 17.4
  Baseline up to Week 76 | 23.2

3. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia for the One-Step and Two-Step Titration Arms During 24-Week Treatment Period
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose less than 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose of study drug at Week 24 or early withdrawal
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Lixisenatide (Two-step Titration): 2-step initiation regimen of lixisenatide.
- Lixisenatide (One-step Titration): 1-step initiation regimen of lixisenatide.
Arm/Group | Lixisenatide (Two-step Titration) | Lixisenatide (One-step Titration)
Number analyzed (Participants) | 33 | 36
participants
  Symptomatic Hypoglycemia | 2 | 1
  Severe Symptomatic Hypoglycemia | 0 | 0

4. Secondary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) for All Patients at Week 52 and 76
Description: Absolute change = HbA1c value at week of assessment (Week 52/Week 76) minus HbA1c value at baseline. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 52, 76
Population: mITT population. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period and "n" = patients with HbA1c assessment for the specified category. Analysis was done on the overall group (pooled data from the 2-step and 1-step titration arms) as pre-specified
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Lixisenatide (Combined)
Number analyzed (Participants) | 47
percentage of hemoglobin
  Week 52 (n=47, observed cases) | -0.83 (0.96)
  Week 76 (n=33, observed cases) | -0.72 (1.20)

5. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 52 and 76
Description: The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Week 52, 76
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide (Combined)
Number analyzed (Participants) | 47
percentage of participants
  Week 52 (n=47, observed cases) | 40.4
  Week 76 (n=33, observed cases) | 27.3

6. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 52 and 76
Description: as for outcome 5
Time Frame: Week 52, 76
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide (Combined)
Number analyzed (Participants) | 47
percentage of participants
  Week 52 (n=47, observed cases) | 14.9
  Week 76 (n=33, observed cases) | 18.2

7. Primary Outcome: Overview of Adverse Event Profile (Treatment Emergent Adverse Events) of the One-Step and Two-Step Titration Arms Assessed Through Adverse Events Collection and Vital Signs, Electrocardiogram (ECG) and Laboratory Monitoring
Description: Overview of adverse event profile is reported in terms of percentage of patients with treatment emergent adverse events (TEAEs) during the 24-week treatment period: any TEAE; any serious TEAE; any TEAE leading to death; and any TEAE leading to permanent treatment discontinuation.
Time Frame: First dose of study drug up to 3 days after the last dose of study drug at Week 24 or early withdrawal
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide (Two-step Titration) | Lixisenatide (One-step Titration)
Number analyzed (Participants) | 33 | 36
percentage of participants
  Any TEAE | 81.8 | 88.9
  Any Serious TEAE | 6.1 | 0
  Any TEAE Leading to Death | 0 | 0
  Any TEAE Leading to Treatment Discontinuation | 9.1 | 11.1

8. Secondary Outcome: Change From Baseline in Body Weight for All Patients at Week 52 and 76
Description: Change was calculated by subtracting baseline value from value at week of assessment (Week 52/Week 76). The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 52, 76
Population: mITT population. Number of patients analyzed=patients with baseline and at least 1 post-baseline weight assessment during on-treatment period and "n" = patients with weight assessment for the specified category. Analysis was done on the overall group (pooled data from the 2-step and 1-step titration arms) as pre-specified
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Lixisenatide (Combined)
Number analyzed (Participants) | 47
kilogram
  Week 52 (n=47, observed cases) | -1.67 (2.10)
  Week 76 (n=33, observed cases) | -1.58 (2.15)

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) for All Patients at Week 52 and 76
Description: Change was calculated by subtracting baseline value from value at week of assessment (Week 52/Week 76). The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 1 day after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 52, 76
Population: mITT population. Number of patients analyzed=patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period and "n" = patients with FPG assessment for the specified category. Analysis was done on the overall group (pooled data from the 2-step and 1-step titration arms) as pre-specified
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lixisenatide (Combined)
Number analyzed (Participants) | 47
mmol/L
  Week 52 (n=47, observed cases) | -0.96 (1.54)
  Week 76 (n=33, observed cases) | -0.46 (2.08)

10. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia for All Patients During On-Treatment Period
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose less than 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.The on-treatment period was the time from the first dose of study drug up to 3 days after the last dose.
Time Frame: First dose of study drug up to 3 days after the last dose of study drug at Week 76 or early withdrawal
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lixisenatide (Combined)
Number analyzed (Participants) | 69
participants
  Symptomatic hypoglycemia | 5
  Severe symptomatic hypoglycemia | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration up to week 76
Description: Median exposure to study treatment was 531 and 533 days in lixisenatide two-step titration and lixisenatide one-step titration arms, respectively. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Arm/Group | Lixisenatide (Two-step Titration) | Lixisenatide (One-step Titration)
Serious Adverse Events (participants affected / at risk) | 2/33 | 1/36
Other Adverse Events (participants affected / at risk) | 24/33 | 34/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (Two-step Titration) (N=33) | Lixisenatide (One-step Titration) (N=36)
Gastroenteritis (Infections and infestations) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (Two-step Titration) (N=33) | Lixisenatide (One-step Titration) (N=36)
Nasopharyngitis (Infections and infestations) | 9 | 13
Pharyngitis (Infections and infestations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 6 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 2 — Hypoglycaemia adverse event is based on investigator reported hypoglycaemia.
Headache (Nervous system disorders) | 0 | 2
Diabetic retinopathy (Eye disorders) | 2 | 1
Yawning (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 5 | 6
Abdominal distension (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 3
Dental caries (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 12 | 18
Toothache (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 2
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Early satiety (General disorders) | 1 | 4
Fatigue (General disorders) | 2 | 2
Neutrophil count decreased (Investigations) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.